CLINICAL TRIAL: NCT05469802
Title: A Randomized, Observer-Blind, Placebo-Controlled, Phase 2 Trial to Evaluate the Safety and Immunogenicity of the Purified Inactivated Zika Virus Vaccine (PIZV) Administered on Days 1 and 29 in Healthy Participants Aged 18 to 49 Years in the US
Brief Title: A Study of Purified Inactivated Zika Virus Vaccine (PIZV) in Healthy Adults
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Business reason, change in Zika virus epidemiology
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ZIK-201
Record Dates: First submitted 2022-07-20; First posted 2022-07-22 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Healthy Volunteers
Keywords: Drug Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- PIZV 0.5 mL (Experimental): Participants will receive PIZV 0.5 mL injection, IM, once on Day 1 (first dose) and Day 29 (second dose).
  Interventions: Biological: Purified Inactivated Zika Virus Vaccine (PIZV)
- Placebo 0.5 mL (Placebo Comparator): Participants will receive a placebo injection, IM, once on Day 1 (first dose) and Day 29 (second dose).
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Purified Inactivated Zika Virus Vaccine (PIZV) — PIZV vaccine with aluminium hydroxide adjuvant IM injection.
  Other Names: TAK-426
  Arms: PIZV 0.5 mL
Other: Placebo — Placebo (normal saline (0.9% NaCl) IM injection.
  Arms: Placebo 0.5 mL

SUMMARY:
The purpose of this study is to describe the side effects and immune response of a candidate vaccine that might protect against Zika. The vaccine called PIZV (purified inactivated Zika virus vaccine) is given by injection in two doses that are 28 days apart in healthy adults. Participants will receive PIZV or placebo and will be followed for 7 days after each dose and up to 6 months after dose 2.

DETAILED DESCRIPTION:
The candidate vaccine being tested in this study is called PIZV (purified inactivated zika virus vaccine) or TAK-426. This study will look at the safety and immunogenicity of PIZV in healthy participants.

The study will enroll approximately 78 healthy participants (≥18 to 49 years) following a 2-dose vaccination schedule. Participants will be randomly assigned (by chance, like flipping a coin) in a 2:1 ratio to either PIZV or placebo which will remain undisclosed to the study observer during the study:

* PIZV
* Placebo

Participants will receive PIZV or placebo 0.5 mL intramuscular (IM) injection into the middle third of the deltoid muscle, preferably in the non-dominant arm on Days 1 (Visit 1) and 29 (Visit 3). The seropositivity rate, seroconversion rate, and geometric-mean titers will be measured 28 days post dose 2. Solicited local reactions and systemic adverse events (AEs) will be assessed for 7 days after each vaccination. Unsolicited AEs will be assessed for 28 days after each vaccination and serious AEs (SAEs), AEs of special interest (AESIs), medically-attended AEs (MAAEs), and AEs leading to withdrawal from the trial throughout the entire study period.

This multi-center trial will be conducted in the United States (US). Trial participants will be in this study for 7 months.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy participants.
2. Participants who can comply with trial procedures (including new trial technologies) and are available for the duration of follow-up.
3. All females of childbearing potential must have a negative urine beta human chorionic gonadotropin (β-hCG) pregnancy test prior to receiving any dose.

Exclusion Criteria:

1. Participants with past or current ZIKV infection by self-report.
2. Participants with past or current dengue virus, yellow fever virus, Japanese encephalitis virus, tick-borne encephalitis virus or West Nile virus infection by self-report.

   Participants who have travelled to dengue and/or Zika endemic countries and US regions and territories*, or who plan to travel to these countries/regions within 1 month prior to anticipated enrollment up to 1 month post dose 2.

   *Centers for Disease Control and Prevention (CDC) website describes dengue/Zika endemic countries and US regions and territories.
3. Participants with any history of progressive or severe neurologic disorder, seizure disorder or neuro-inflammatory disease (e.g., Guillain-Barré syndrome).
4. Participants with known or suspected impairment/alteration of immune function, including:

   1. Chronic use of oral or parenteral steroids (equivalent to 20 mg/day prednisone ≥12 weeks / ≥2 mg/kg body weight/day prednisone ≥2 weeks) within 60 days prior to Day 1 (use of inhaled, intranasal, or topical corticosteroids is allowed).
   2. Receipt of immunomodulatory agents within 60 days prior to Day 1.
   3. Receipt of parenteral, epidural or intra-articular immunoglobulin preparation, blood products, and/or plasma derived products within 3 months prior to Day 1 or planned receipt during the full length of the trial. In addition, participants must be advised not to donate blood during the study period.
   4. Known Human Immunodeficiency Virus (HIV) infection or HIV-related disease.
   5. Genetic immunodeficiency.
5. Participants with known current or chronic hepatitis B and/or hepatitis C infections.
6. Participants with abnormalities of splenic or thymic function.
7. Participants with a known bleeding diathesis, or any condition that may be associated with a prolonged bleeding time.
8. Participants with any serious chronic or progressive disease according to the judgment of the investigator (e.g., neoplasm, insulin-dependent diabetes, cardiac, renal, hepatic or thyroid disease, uncontrolled hypertension, uncontrolled asthma).
9. Participants with a history of substance or alcohol abuse within the past 2 years.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2024-01-02 (Estimated); Primary Completion 2024-07-05 (Estimated); Study Completion 2024-07-05 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Seropositivity for Neutralizing Antibodies Against Zika Virus at 28 Days Post Dose 2 | Within 28 days after Dose 2 (Day 57)
  Seropositive participants are defined as participants with quantifiable (tested positive at or above the limit of quantitation [LOQ]) serum neutralizing anti-Zika virus (ZIKV) antibodies. Data will be reported for the overall study population (regardless of pre-vaccination flavivirus (FV) serostatus) and in FV naïve participants only.
Percentage of Participants With Seroconversion for Neutralizing Antibodies Against Zika Virus at 28 Days Post Dose 2 | Within 28 days after Dose 2 (Day 57)
  Seroconversion is defined as the percentage of participants with either pre-vaccination titer <LOQ and a post-vaccination titer ≥4xLOQ; or a pre-vaccination titer ≥LOQ and a 4-fold increase in titer post vaccination. Data will be reported for the overall study population (regardless of pre-vaccination FV serostatus) and in FV naïve participants only.
Geometric Mean Titers (GMTs) for Neutralizing Antibodies Against Zika Virus at 28 Days Post Dose 2 | Within 28 days after Dose 2 (Day 57)
  GMTs for neutralizing antibodies against ZIKV will be measured by assessing the quantity of neutralizing antibodies that bind ZIKV. Data will be reported for the overall study population (regardless of pre-vaccination FV serostatus) and in FV naïve participants only.
Percentage of Participants With Solicited Local Injection Site Reactions for 7 Days After First Dose of Vaccination | Within 7 days after Dose 1 (Up to Day 7)
  Solicited local AEs (at injection site) included pain/tenderness (mild: mild discomfort to touch, moderate: discomfort with movement, severe: significant discomfort at rest, potentially life-threatening: emergency room [ER] visit or hospitalization), erythema/redness (mild: 2.5 - 5 cm, moderate: 5.1 - 10 cm, severe: > 10 cm, potentially life-threatening: necrosis or exfoliative dermatitis), and swelling/induration (mild: 2.5 - 5 cm and does not interfere with activity, moderate: 5.1 - 10 cm or interferes with activity, severe: > 10 cm or prevents daily activity, potentially life-threatening: Necrosis). Data will be reported for the overall study population and in FV naïve participants only.
Percentage of Participants With Solicited Local Injection Site Reactions for 7 Days After Second Dose of Vaccination | Within 7 days After Dose 2 (Days 29 to 35)
  Solicited local AEs (at injection site) included pain/tenderness (mild: mild discomfort to touch, moderate: discomfort with movement, severe: significant discomfort at rest, potentially life-threatening: ER visit or hospitalization), erythema/redness (mild: 2.5 - 5 cm, moderate: 5.1 - 10 cm, severe: > 10 cm, potentially life-threatening: necrosis or exfoliative dermatitis), and swelling/induration (mild: 2.5 - 5 cm and does not interfere with activity, moderate: 5.1 - 10 cm or interferes with activity, severe: > 10 cm or prevents daily activity, potentially life-threatening: Necrosis). Data will be reported for the overall study population and in FV naïve participants only.
Percentage of Participants With Solicited Systemic Adverse Events (AEs) for 7 Days After First Dose of Vaccination | Within 7 days after Dose 1 (Up to Day 7)
  Solicited systemic AEs included fever, headache, fatigue, malaise, arthralgia, and myalgia that occurred within 7 days of first vaccination. Solicited systemic AEs will be graded from 1(mild) to 4(potentially life threatening) by severity. Fever: Grade 1(mild)= 38.0-38.4 degrees Celsius(°C)/100.4-101.1 degrees Fahrenheit (°F), Grade 2(moderate)=38.5-38.9°C/101.2-102.0°F, Grade 3(severe)=39.0-40°C/102.1-104°F, Grade 4 (potentially life threatening)=>40°C/>104°F. Headache, fatigue, malaise, arthralgia, and myalgia: Grade 1=no interference with activity, Grade 2=some interference with activity(Headache: repeated use of non-narcotic pain reliever>24 hours or some interference with activity), Grade 3 =significant; prevents daily activity(Headache: significant; any use of narcotic pain reliever or prevents daily activity), and Grade 4=ER visit or hospitalization. Data will be reported for the overall study population and in FV naïve participants only.
Percentage of Participants With Solicited Systemic AEs for 7 Days After Second Dose of Vaccination | Within 7 days After Dose 2 (Days 29 to 35)
  Solicited systemic AEs included fever, headache, fatigue, malaise, arthralgia, and myalgia that occurred within 7 days of first vaccination. Solicited systemic AEs will be graded from 1(mild) to 4(potentially life threatening) by severity. Fever: Grade 1(mild)= 38.0-38.4°C/100.4-101.1°F, Grade 2(moderate)=38.5-38.9°C/101.2-102.0°F, Grade 3(severe)=39.0-40°C/102.1-104°F, Grade 4 (potentially life threatening)=>40°C/>104°F. Headache, fatigue, malaise, arthralgia, and myalgia: Grade 1=no interference with activity, Grade 2=some interference with activity(Headache: repeated use of non-narcotic pain reliever>24 hours or some interference with activity), Grade 3 =significant; prevents daily activity(Headache: significant; any use of narcotic pain reliever or prevents daily activity), and Grade 4=ER visit or hospitalization. Data will be reported for the overall study population and in FV naïve participants only.
Percentage of Participants With at Least One Unsolicited AE for 28 Days After First Dose of Vaccination | Within 28 days after dose 1 (Up to Day 29)
  An unsolicited AE is any AE reported by the participant that is either not specified as a solicited AE or is specified as a solicited AE but starts outside the period for reporting solicited AE (ie, 7 days in total including the day of PIZV or placebo administration). Unsolicited AEs will be graded from 1 to 4 by severity, where Grade 1 (mild)= no interference with activity, Grade 2 (moderate)= some interference with activity, Grade 3 (severe)= significant; prevents daily activity, and Grade 4 (potentially life threatening)= ER visit or hospitalization. Data will be reported for the overall study population and in FV naïve participants only.
Percentage of Participants With at Least One Unsolicited AE for 28 Days After Second Dose of Vaccination | Within 28 days after dose 2 (Days 29 to 57)
  An unsolicited AE is any AE reported by the participant that is either not specified as a solicited AE or is specified as a solicited AE but starts outside the period for reporting solicited AE (ie, 7 days in total including the day of PIZV or placebo administration). Unsolicited AEs will be graded from 1 to 4 by severity, where Grade 1 (mild)= no interference with activity, Grade 2 (moderate)= some interference with activity, Grade 3 (severe)= significant; prevents daily activity, and Grade 4 (potentially life threatening)= ER visit or hospitalization. Data will be reported for the overall study population and in FV naïve participants only.
Percentage of Participants With at Least One Serious Adverse Event (SAE) Throughout the Entire Study Period | From day of first vaccination (Day 1) up to end of the study (Day 211)
  An SAE will be defined as any untoward medical occurrence that: 1) results in death, 2) is life-threatening, 3) requires inpatient hospitalization or prolongation of existing hospitalization, 4) results in persistent or significant disability/incapacity, 5) leads to a congenital anomaly/birth defect in the offspring of the participant or 6) is an important medical event that satisfies any of the following: a) May require intervention to prevent items 1 through 5 above. b) May expose the participant to danger, even though the event is not immediately life threatening or fatal or does not result in hospitalization. Data will be reported for the overall study population and in FV naïve participants only.
Percentage of Participants With at Least One Adverse Events of Special Interest (AESI) Throughout the Entire Study Period | From day of first vaccination (Day 1) up to end of the study (Day 211)
  An AE is defined as any untoward medical occurrence in a clinical investigation participant administered an PIZV or placebo; it does not necessarily have to have a causal relationship with PIZV or placebo administration. AESI is defined as an AE collected through the study period and entered in the eCRF by the investigator or designee within 24 hours of becoming aware of the event which includes new onset of or worsening of the following neurologic diseases: Guillain-Barré syndrome (GBS), acute disseminated encephalomyelitis, idiopathic peripheral facial nerve palsy (Bell's palsy), seizures including but not limited to febrile seizures and/or generalized seizures/convulsions, and anaphylaxis. Data will be reported for the overall study population and in FV naïve participants only.
Percentage of Participants With at Least One Medically-Attended Adverse Event (MAAE) Throughout the Entire Study Period | From day of first vaccination (Day 1) up to end of the study (Day 211)
  AE: any untoward medical occurrence in a clinical investigation participant administered PIZV or placebo; it does not necessarily have to have a causal relationship with trial vaccine administration. MAAEs is defined as AEs leading to an unscheduled visit to or by a healthcare professional including visits to an emergency department, but not fulfilling seriousness criteria. Data will be reported for the overall study population and in FV naïve participants only.

SECONDARY OUTCOMES:
Percentage of Participants With Seropositivity for Neutralizing Antibodies Against Zika Virus | Within 28 days after Dose 1 (Day 29) and 6 months after Dose 2 (Day 211)
  Seropositive participants are defined as participants with quantifiable (tested positive at or above the LOQ) serum neutralizing anti-ZIKV antibodies. Data will be reported for the overall study population and in FV naïve participants only.
Percentage of Participants With Seropositivity for Neutralizing Antibodies Against Zika Virus in FV Exposed Participants | Baseline (Day 1), within 28 days after Dose 1 (Day 29), 28 days after Dose 2 (Day 57) and 6 months after Dose 2 (Day 211)
  Seropositive participants are defined as participants with quantifiable (tested positive at or above the LOQ) serum neutralizing anti-ZIKV antibodies. Data will be reported for FV exposed participants only.
Percentage of Participants With Seroconversion for Neutralizing Antibodies Against Zika Virus | Within 28 days after Dose 1 (Day 29) and 6 months after Dose 2 (Day 211)
  Seroconversion is defined as the percentage of participants with either pre-vaccination titer <LOQ and a post-vaccination titer ≥4xLOQ; or a pre-vaccination titer ≥LOQ and a 4-fold increase in titer post vaccination. Data will be reported for the overall study population and in FV naïve participants only.
Percentage of Participants With Seroconversion for Neutralizing Antibodies Against Zika Virus in FV Exposed Participants | Within 28 days after Dose 1 (Day 29), 28 days after Dose 2 (Day 57) and 6 months after Dose 2 (Day 211)
  Seroconversion is defined as the percentage of participants with either pre-vaccination titer <LOQ and a post-vaccination titer ≥4xLOQ; or a pre-vaccination titer ≥LOQ and a 4-fold increase in titer post vaccination. Data will be reported for FV exposed participants only.
Geometric Mean Titers (GMTs) for Neutralizing Antibodies Against Zika Virus | Baseline (Day 1), within 28 days after Dose 1 (Day 29) and 6 months after Dose 2 (Day 211)
  GMTs for neutralizing antibodies against ZIKV will be measured by assessing the quantity of neutralizing antibodies that bind ZIKV. Data will be reported for the overall study population and in FV naïve participants only.
GMTs for Neutralizing Antibodies Against Zika Virus in FV Exposed Participants | Baseline (Day 1), within 28 days after Dose 1 (Day 29), 28 days after Dose 2 (Day 57) and 6 months after Dose 2 (Day 211)
  GMTs for neutralizing antibodies against ZIKV will be measured by assessing the quantity of neutralizing antibodies that bind ZIKV. Data will be reported for FV exposed participants only.
Percentage of Participants With at Least One Serious Adverse Event (SAE) From 28 Days up to 6 Months Post Dose 2 | From 28 days up to 6 months post Dose 2 (Up to Day 211)
  An SAE will be defined as any untoward medical occurrence that: 1) results in death, 2) is life-threatening, 3) requires inpatient hospitalization or prolongation of existing hospitalization, 4) results in persistent or significant disability/incapacity, 5) leads to a congenital anomaly/birth defect in the offspring of the participant or 6) is an important medical event that satisfies any of the following: a) May require intervention to prevent items 1 through 5 above. b) May expose the participant to danger, even though the event is not immediately life threatening or fatal or does not result in hospitalization. Data will be reported for the overall study population and in FV naïve participants only.
Percentage of Participants With at Least One SAE in FV Exposed Participants | Within 28 days post Dose 1 (Day 29), 28 days post Dose 2 (Day 57) and 6 months post Dose 2 (Up to Day 211)
  An SAE will be defined as any untoward medical occurrence that: 1) results in death, 2) is life-threatening, 3) requires inpatient hospitalization or prolongation of existing hospitalization, 4) results in persistent or significant disability/incapacity, 5) leads to a congenital anomaly/birth defect in the offspring of the participant or 6) is an important medical event that satisfies any of the following: a) May require intervention to prevent items 1 through 5 above. b) May expose the participant to danger, even though the event is not immediately life threatening or fatal or does not result in hospitalization. Data will be reported for FV exposed participants only.
Percentage of Participants With at Least One Adverse Events of Special Interest (AESI) From 28 Days up to 6 Months Post Dose 2 | From 28 days up to 6 months post Dose 2 (Up to Day 211)
  AE: any untoward medical occurrence in a clinical investigation participant administered PIZV or placebo; it does not necessarily have to have a causal relationship with trial vaccine administration. An AE will be considered AESI if any participant experiences a new onset of or worsening of the following neurologic diseases: GBS, acute disseminated encephalomyelitis, idiopathic peripheral facial nerve palsy (Bell's palsy), seizures including but not limited to febrile seizures and/or generalized seizures/convulsions and/or anaphylaxis. Data will be reported for the overall study population and in FV naïve participants only.
Percentage of Participants With at Least One AESI in FV Exposed Participants | Within 28 days post Dose 1 (Day 29), 28 days post Dose 2 (Day 57) and 6 months post Dose 2 (Up to Day 211)
  AE: any untoward medical occurrence in a clinical investigation participant administered PIZV or placebo; it does not necessarily have to have a causal relationship with trial vaccine administration. An AE will be considered AESI if any participant experiences a new onset of or worsening of the following neurologic diseases: GBS, acute disseminated encephalomyelitis, idiopathic peripheral facial nerve palsy (Bell's palsy), seizures including but not limited to febrile seizures and/or generalized seizures/convulsions and/or anaphylaxis. Data will be reported for FV exposed participants only.
Percentage of Participants With at Least One Medically-Attended Adverse Event (MAAE) From 28 Days up to 6 Months Post Dose 2 | From 28 days up to 6 months post Dose 2 (Up to Day 211)
  AE: any untoward medical occurrence in a clinical investigation participant administered PIZV or placebo; it does not necessarily have to have a causal relationship with trial vaccine administration. MAAEs is defined as AEs leading to an unscheduled visit to or by a healthcare professional including visits to an emergency department, but not fulfilling seriousness criteria. Data will be reported for the overall study population and in FV naïve participants only.
Percentage of Participants With at Least One MAAE in FV Exposed Participants | Within 28 days post Dose 1 (Day 29), 28 days post Dose 2 (Day 57) and 6 months post Dose 2 (Up to Day 211)
  AE: any untoward medical occurrence in a clinical investigation participant administered PIZV or placebo; it does not necessarily have to have a causal relationship with trial vaccine administration. MAAEs is defined as AEs leading to an unscheduled visit to or by a healthcare professional including visits to an emergency department, but not fulfilling seriousness criteria. Data will be reported for FV exposed participants only.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (5):
- United States (5):
  - CenExel Research Centers of America, Oakland Park, Florida
  - Velocity Clinical Research, Boise, Meridian, Idaho
  - AMR East Wichita, Formerly Heartland Associates East Wichita, an AMR company, Wichita, Kansas
  - AMR Lexington, Formerly Central Kentucky Research Associates, an AMR company, Lexington, Kentucky
  - Alliance for Multispecialty Research, LLC, Kansas City, Missouri

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information about this study, click this link. — https://clinicaltrials.takeda.com/study-detail/959a893ca7334342?idFilter=%5B%22ZIK-201%22%5D